CLINICAL TRIAL: NCT00004275
Title: Phase II Randomized Study of Oxandrolone vs Placebo for Growth Hormone-Treated Girls With Turner's Syndrome
Brief Title: Oxandrolone Compared With a Placebo on Growth Rate in Girls With Growth Hormone-Treated Turner's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Jefferson Medical College of Thomas Jefferson University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11681; TJU-11681
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Turner's Syndrome
Keywords: Turner's syndrome; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Turner Syndrome; Genetic Diseases, Inborn; Rare Diseases | interventions — Growth Hormone; Oxandrolone

INTERVENTIONS:
Drug: growth hormone
Drug: oxandrolone

SUMMARY:
RATIONALE: Turner's syndrome is a disease in which females are missing all or part of one X chromosome and do not produce the hormones estrogen and androgen. Giving growth hormone may help girls with Turner's syndrome attain a more normal height. It is not yet known if growth hormone is more effective with or without oxandrolone for Turner's syndrome.

PURPOSE: Randomized phase II trial to study the effectiveness of oxandrolone in girls who have growth hormone-treated Turner's syndrome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are randomly assigned to recombinant human growth hormone (GH) and oxandrolone versus GH and placebo.

GH is administered by daily subcutaneous injection and oxandrolone is given every day by mouth. Treatment continues for 3 years; estrogen is offered after year 2.

A study duration of 8 years is anticipated.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Turner's syndrome-compatible karyotype No Y material in peripheral karyotype Bone age no greater than 11 years --Prior/Concurrent Therapy-- No more than 12 months of prior estrogen, androgen, or growth hormone

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80
Dates: Start 1999-10; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Ross, Study Chair — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Jefferson Medical College of Thomas Jefferson University, Philadelphia, Pennsylvania, United States